CLINICAL TRIAL: NCT05866835
Title: Validation of a Generic Procedure for the Fabrication of a Custom-made Intra-oral Protection Using an Inter-arch Piece
Brief Title: Validation of a Digitalised Intraoral Protection
Acronym: NUPPIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/61
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ventilatory Performances of Athletes During the Use of the Intra-oral Protections
Keywords: ventilatory performance; athlete; intra-oral protection; protection
MeSH Terms: interventions — Pulmonary Ventilation

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Athlete (Experimental): healthy, adult or minor (16 years or older), high-level sportsmen and women, volunteers
  Interventions: Other: Manufacture of custom-made IOP; Other: Ventilation tests; Other: Evaluation of comfort level:

INTERVENTIONS:
Other: Manufacture of custom-made IOP — Manufacture of custom-made "unimaxillary" and "modified unimaxillary" intra-oral protection (IOP) with vertical dimensions of 4 mm and 6 mm. 3D modeling of a IOP based on:
  * digital recording of the maxillary and mandibular dental arches
  * mandibular wedging performed with an inter-arch piece
  * digital recording of the inter-arch position
Other: Ventilation tests — Realization of a ventilation test (VO2max) to determine the Maximum Aerobic Speed (MAS).
  Measurement of ventilatory parameters without IOP and with each IOP :
  * At rest, standing still.
  * During a 4 minute run on a treadmill at 50% of MAS.
  * During a 4-minute run on a treadmill, at a speed corresponding to 70% of MAS
Other: Evaluation of comfort level: — Collection from participants (self-questionnaire)

SUMMARY:
Type III (custom-made) intra-oral protection (IOP) models represent 13% of IOP worn by amateur rugby club players in France.

However, this model is recognized as the most effective when made in accordance with essential health and safety requirements.

This observation is at the origin of a new approach that the investigators are proposing with the objective of removing the barriers to access to custom-made IOP. This research is based on the combination of new digital technologies, scanning and 3D printing, to develop a new generation of IOP.

This project aims to show the interest of this new generation of "modified unimaxillary" IOP on the ventilation of the athletes and his/her comfort when he/she evolves with his IOP in place

DETAILED DESCRIPTION:
Type III (custom) Intra Oral Protection (IOP) models represent 13% of IOP worn by amateur rugby players in France.

However, this model is recognized as the most effective when made in accordance with essential health and safety requirements.

This under-utilization can be explained by the existence of many barriers to the diffusion of custom-made IOP:

1. Organizational barrier: long fabrication procedure (minimum 3 sessions) requiring qualified people (dental surgeon, dental technician), trained in the technique of making custom IOP and in essential health and safety criteria.
2. Financial barrier: high cost with a selling price of 200€ to 300€ per unit.
3. Technical barriers:

   * Difficulties in making custom-made IOP for athletes who wear fixed braces (brackets and wire),
   * Difficulties in improving the impact energy dissipation capacity without affecting the absorption capacity of the custom-made IOP,
   * Difficulties in individualizing and characterizing the IOP.

This observation is at the origin of a new approach proposed in order to remove the barriers to access to custom IOP. Naturally, this project relies on the combination of new digital technologies, scanning and 3D printing, to develop a new generation IOP with :

* A simpler and shorter procedure,
* A target price accepted by athletes,
* "French Association for Standardization"(AFNOR) standards guaranteed,
* Compatibility with fixed orthodontic treatments,
* Ability to develop new protection strategies,
* Ability to improve the athlete's comfort. Currently, the IOP resulting from these technologies are mainly "unimaxillary", i.e. without engagement of the mandibular dental arch and without ventilation space. In order to comply with the Afnor XP S72-427 standard, the project proposes the fabrication of two models of "modified unimaxillary" IOP that ensure the engagement of the mandibular dental arch and the creation of a ventilation space at two different heights, 4mm and 6mm. This project aims to show the interest of this new generation of "modified unimaxillary" IOP on the athlete's ventilation and his comfort when he evolves with his IOP in place. It is based on a population of men and women, minors and adults, practicing a sport at risk of oral trauma and uses a methodology already proven by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 16 and 35,
* Subject affiliated to a social security system,
* Subject affiliated with the French Federation of Boxing or Rugby or Football
* Subject having signed a consent form
* For minors, legal guardians having signed the free and informed consent form

Exclusion Criteria:

* Subject with a pathology incompatible with the realization of the trial:

  * Absolute contraindications: Recent infarction (wait 5 to 12 days depending on severity), Threat syndrome (lawful test after stabilization - at least 3 days without spontaneous seizures), Resting BP > 200/120 mmHg, Uncompensated heart failure, Third-degree Atrioventricular block, Myocarditis, Pericarditis, Endocarditis, Aortic Dissection, Intracardiac tumor or thrombus, Deep venous thrombosis, Pulmonary Embolism,
  * Relative contraindications: Aortic stenosis (formal contraindication if lipothymia, syncope or signs of heart failure), Severe non-revascularized coronary artery disease, Pulmonary arterial hypertension (formal contraindication if primary), Severe rapid ventricular or supraventricular arrhythmias
* Subject under B-mimetic drug treatment,
* Subject with decaying teeth,
* Subject under court protection,
* Subject participating in another research study,
* Subject in pregnancy.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Ventilatory flow per minute | 3 weeks (W3) after inclusion (W0)
  The ventilatory flow rate per minute will be measured during the ventilation test

SECONDARY OUTCOMES:
Confort level | 3 weeks (W3) after inclusion (W0)
  For the evaluation of the comfort level of wearing the IOP, eleven judgement criteria are proposed and evaluated using a visual analogue scale graduated from 0 (uncomfortable) to 10 (very comfortable): retention, muco-gingival aspect, height of mouth opening, volume of the PIB, nausea, phonation, open mouth ventilation, clenched jaw ventilation, salivation, masticatory muscles, temporomandibular joint.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CREPS de Bordeaux, Bordeaux
  - Institut national du sport, de l'expertise et de la performance (INSEP), Paris